CLINICAL TRIAL: NCT06711601
Title: Ultrasound Evaluation Of Two Anatomic Landmarks In Spinal Anesthesia For Cesarean Section: The Posterior Superior Iliac Spine vs Iliac Crest
Acronym: USPSISICL
Status: Recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: [2024] No. 131
Record Dates: First submitted 2024-11-18; First posted 2024-12-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Spinal Anesthesia; Ultrasonography; Posterior Superior Iliac Spine; Intercristal Line
Keywords: cesarean section; ultrasonography; spinal anesthesia; Posterior Superior Iliac Spine; intercristal line

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T group: The intercristal line-based palpation protocol followed the rule described by Kim et al[19], with minor modifications to accommodate the flexed lateral decubitus position: Select the interspinous space that is either intersected by the intercristal line or lies immediately below it.
- P group: The PSIS line-based palpation protocol stipulated targeting the L3/4 interspinous space within the an interval using hierarchical rules: single spaces are labeled L3/4; for two spaces, L3/4 is the intercristal line-intersected one (or lower if neither); for rare three spaces, the lowest is L3/4
- Group M: Based on an interim analysis of Phase 1 data, we established the following decision protocol for L3/4 interspinous space localization:
  1. PI ≥9 cm: Select the interspace at or immediately below the PI line.
  2. PI ≤7 cm: Select the interspace at or immediately above the PI line.
  3. PI 7-9 cm: Apply a 6.5-10 cm target window from the PSIS point.
     * If one interspace lies within this window, select it.
     * If multiple interspaces are present, choose the most caudal one.

SUMMARY:
Intercristal line as palpation landmarks to identifying the vertebral level is frequently inaccurate.To find more safe and reliable body surface markers and convenient methods to be solved in clinical work.The investigators performed a two-stage study to evaluated the accuracy of intercristal line and the The Posterior Superior Iliac Spine (PSIS) line to identify the lumbar interspinous spaces for spinal anesthesia using ultrasonography in pregnant woman which will provide a second option.

DETAILED DESCRIPTION:
The investigators performed a two-stage study to evaluated the accuracy of Intercristal line and the PSIS line to identify the lumbar intervertebral space for spinal anesthesia using ultrasonography in pregnant woman. In phase 1, the distances between the PSIS line and each lumbar interspinous space is measured by ultrasound,and the mean and 95% confidence interval of distances in pregnant women with different height ranges were calculated to provide a reference for identifying specific lumbar spaces.In phase 2, a further 230 participants were received the PSIS, Intercristal line or both as palpation landmarks to define specific lumbar spaces.

ELIGIBILITY:
Inclusion Criteria:

* After obtaining written informed consents,pregnant women at 37-42 weeks of gestation

Exclusion Criteria:

* BMI ≥ 40 kg/m² (to minimize palpation variability), History of lumbar surgery/deformity (scoliosis, spondylolisthesis or osteoporotic vertebral collapse), Inability to maintain the flexed lateral decubitus position, Participant withdrawal, Unforeseen anatomical anomalies discovered during screening.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We enrolled parturients aged 22-45 years at 37-42 weeks of gestation scheduled for epidural or combined spinal-epidural anesthesia (for labor or cesarean section)
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
The distance between the PSIS line and each mid-interspinous space | three days
  PSIS line was defined as an intercristal line drawn between the the final posterior superior iliac spine point.Use a ruler to measure the distance between the PSIS line and each midddle- interspinous space （L1/2 through L5/S1）and record. The mean of distances and 95% confidence interval are calculated.
The accuracy of the anatomic landmarks to determine the L3/4 interspinous space | three days
  The L3-L4 intervertebral space was detected using intercristal line and the PSIS line in a random order by 2 experienced anesthesiologists. After determining the L3-L4 intervertebral space using each method alternately, horizontal skin marks were created with an erasable pen. Then, another experienced anesthesiologist for ultrasonographic examination assessed the intervertebral spaces.After identifying the sacrum, the investigator moved the probe in a cephalad direction, counted the intervertebral spaces and assessed the actual intervertebral spaces of the 2 skin marks.

SECONDARY OUTCOMES:
The distance between the palpated intercristal line and PSIS line | three days
  palpated intercristal line line was identified and marked by bilateral palpation of the iliac crest summits.
  Subsequently, two reference points were defined: "point PSIS" (intersection of the PSIS line with the spinal midline) and "point PI" (intersection of the PI line with the spinal midline). We then calculated the following three distances: the "L3/4 distance" (from the L3/4 interspinous space midpoint to point PSIS), the "PI distance" (from point PI to point PSIS) The experienced anesthesiologist for ultrasonographic examination assessed the actual interspinous space of the intercristal line.
baseline data | three days
  The age
baseline data | three days
  body mass index (BMI)
Maternal height | three days
  Maternal height
baseline data | three days
  waist circumference
baseline data | three days
  the gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Souping Wang, PhD, Study Director — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No